CLINICAL TRIAL: NCT05347901
Title: Clinical Precise Diagnosis and Treatment of Personalized Z-score Evaluation Combined With Genomic Analysis in the Repair of Coronary Artery Injury in Kawasaki Disease
Brief Title: Clinical Precise Diagnosis and Treatment in the Kawasaki Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Children's Hospital of Fudan University Qidong Branch (Unknown); Second Affiliated Hospital of Nantong University (Other); Jiangsu Hai'an People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: LCYJ-A06
Record Dates: First submitted 2022-03-23; First posted 2022-04-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-04

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health Control: Health children with age and sex paired with experimental group
  Interventions: Diagnostic Test: Echocardiography, Genomics NGS sequencing
- Kawasaki Disease: KD patients, with no congenital heart disease, metabolic disease or Immune deficiency disease.
  Interventions: Diagnostic Test: Echocardiography, Genomics NGS sequencing

INTERVENTIONS:
Diagnostic Test: Echocardiography, Genomics NGS sequencing — The inner diameter of left main coronary artery, anterior descending branch, circumflex branch and right coronary artery was measured by echocardiography. Blood samples were send for genomics NGS sequencing

SUMMARY:
The purpose of this project is to explore the differential gene expression profile of Kawasaki disease, and will explore the diagnosis and treatment targets related to coronary artery injury or kawasaki disease susceptibility, vascular damage, IVIG (intravenous immunoglobulin) treatment resistance, incomplete Kawasaki disease, etc.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will acquire blood samples with complete clinical data and prognostic information. Using clinicopathology, molecular biology, gene diagnostics and other techniques to verify the expression differences of target genes and proteins and analyze their expression levels; To analyze the role of target genes and proteins in the occurrence and development of Kawasaki disease and their correlation with the risk of coronary artery injury. In vitro and in vivo KD (Kawasaki Disease) model was used to investigate the role of target genes in Kawasaki disease by gene interference and various molecular biological techniques.

ELIGIBILITY:
Inclusion Criteria:

* Individual patient's medical file data confirmed the diagnosis of KD using diagnostic criteria issued by the American Heart Association in 2017;
* Patients were respond to IVIG treatment;
* the patients aged from 2 months to 14 years old;
* All included patients required to sign an informed consent form.

Exclusion Criteria:

* The patients with severe infections;
* The patients with a history of tuberculosis or recent close contact with tuberculosis;
* The patient vaccinated with live vaccine in 6 months;
* The patients with the application of hormone or other immunosuppressive agents;
* The patients didn"t want to signed informed consent.

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children under the care of consultant in hospital for Kawasaki disease
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Z-score of coronary artery | 2 weeks
  Calculate z-score by using LMS regression form echocardiography data
Z-score of coronary artery | 4 weeks
  Calculate z-score by using LMS regression form echocardiography data
Differential gene profile | 0 week
  Differential expression analysis of NGS sequencing in genomics
Differential gene profile | 1 week after IVIG treatment
  Differential expression analysis of NGS sequencing in genomics

CONTACTS AND LOCATIONS:
Overall Officials: Jianmei Zhao, PhD., Study Chair — Affiliated Hospital of Nantong University
Locations (4):
- China (4):
  - Affiliated Hospital of Nantong University, Nantong, Jangsu
  - Jiangsu Hailan People's Hospital, Haian, Jiangsu
  - Nantong first People's Hospital, Nantong, Jiangsu
  - Children's Hospital of Fudan University Qidong Branch, Qidong, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided